CLINICAL TRIAL: NCT03703921
Title: Neuroimaging of Pain: Changes in Regional Brain Functioning Associated With Amplified Pain and Intensive Treatment
Status: Completed | Type: Observational
Sponsor: Children's Mercy Hospital Kansas City (Other)
Responsible Party: Principal Investigator, Cara Hoffart, DO, Pediatric Rheumatologist, Children's Mercy Hospital Kansas City
Other Study IDs: RAPS_fMRI_001
Record Dates: First submitted 2018-10-02; First posted 2018-10-12 (Actual); Last update posted 2020-08-06 (Actual); Status verified 2020-08

CONDITIONS: Pain, Chronic
Keywords: Intensive interdisciplinary pain treatment; fMRI; fear of pain
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The proposed study will examine how intensive interdisciplinary pain treatment (IIPT, specifically the Rehabilitation for Amplified Pain Syndrome, or RAPS, program at Children's Mercy Hospital) impacts neurofunctional mechanisms of emotional and physical pain processing in patients. There has been recent interest in characterizing the brain regions responsible for processing pain (Wager et al., 2013), but little research has included youth. A better understanding of the physiological mechanisms of pain can lead to better treatment outcomes.

DETAILED DESCRIPTION:
Youth will be scanned before or during the first week of participation in the Rehabilitation for Amplified Pain Syndrome (RAPS) program, and a second time near or just after program completion (typically 3-5 weeks later). One functional MRI task will involve passive viewing of emotional and pain-related images including some that have been widely used in previous neuroimaging research (e.g., the International Affective Picture Set, Human Facial Expressions; alternating positive and negative affect/valence). The other functional MRI task, will involve systematic external application of somatosensory stimulation (pressure) to the hand in alternating blocks. The entire imaging procedure will take approximately an hour. MRI technicians and/or study staff will administer the scanning protocol. Study team will be responsible for the systematic external application of sensory input.

ELIGIBILITY:
Inclusion Criteria:

* Age 13 to 19
* Admitted to the RAPS program for intensive treatment

Exclusion Criteria:

* Inability to participate in imaging due to developmental delay
* Inability or unwillingness to be still during imaging procedures

Ages: 13 Years to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Target study population is youth ages 13-19, regardless of gender, who have been admitted to the RAPS program for intensive treatment. When offered a spot in the RAPS program, patient/parent will be informed about the study and asked if they would like to be contacted to receive more information. Prior to any study procedures, the permission/assent or consent form will be reviewed carefully with the participant (and parent, if applicable).
Sampling Method: Non-Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2018-07-09 (Actual); Primary Completion 2019-10-31 (Actual); Study Completion 2019-10-31 (Actual)

PRIMARY OUTCOMES:
Change in brain response (as measured by fMRI) to viewing images of physical and emotional pain, and experiencing somatosensory simulation to the arm. | Baseline fMRI will be conducted when the participant starts IIPT. A second scan will be conducted at the end of treatment (3-5 weeks later).
  Participants will undergo scanning without intravenous contrast, performed with a 3-Tesla magnetic resonance imaging (MRI) scanner. Structural scan will be completed for spatial normalization and registration with the functional data. Functional scans use blood-oxygen level dependent (BOLD) assessments during active tasks to determine regional brain activation while viewing pictures and experiencing somatosensory stimulation.

SECONDARY OUTCOMES:
Pain Discounting Questionnaire (PDQ) | Pain Discounting Questionnaire (PDQ), will be completed at the beginning of IIPT (same time as fMRI) and 3-5 weeks later or at the end of the IITP (same time as last fMRI.)
  - Pain Discounting Questionnaire (PDQ). This measures the extent to which later rewards (in this case pain relief) lose value related to the delay (being a number of days later). - This was adapted from the 27-item Monetary-Choice Questionnaire. Scoring procedures include calculating the value of k (hyperbolic discount parameter) for small, medium, and large delays. Using the geometric mean of responses allows for a single score if necessary. The values of k ranges from 0-1. - Greater values indicate more delay discounting, or more tendency to value a sooner, smaller reward rather than wait for a later, larger reward. Subscales are not combined.
Fear of Pain Questionnaire (FOPQ), child and parent report | Fear of Pain Questionnaire (FOPQ), child and parent report will be completed at the beginning of IIPT (same time as fMRI) and 3-5 weeks later or at the end of the IITP (same time as last fMRI.)
  - Fear of Pain Questionnaire, child report (FOPQ-C) and Fear of Pain Questionnaire, parent proxy report (FOPQ-P). These each measures the extent to which youth with chronic pain experience cognitive and physiological signs of fear when experiencing pain. Scale ranges: - FOPQ-C total: 24 items, range 0-96, FOPQ-C fear of pain: 13 items, range 0-52, FOPQ-C avoidance of activities: 11 items, range 0-44, FOPQ-P total: 21 items, range 0-84, FOPQ-P fear of pain: 8 items, range 0-32, FOPQ-P avoidance of activities: 10 items, range 0-40, FOPQ-P school avoidance: 5 items, range 0-20. For all total scores and subscales, greater scores indicate more fear of pain. For both the FOPQ-C and FOPQ-P, the total scores indicate a sum of all items.

CONTACTS AND LOCATIONS:
Locations (1):
- Children's Mercy Hospital, Kansas City, Missouri, United States

IPD SHARING:
Plan to Share IPD: No
Individual data will be retained at our institution.